CLINICAL TRIAL: NCT02238795
Title: Sepsis-Associated Purpura Fulminans International Registry - Europe
Acronym: SAPFIRE
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Medical University of Vienna (Other); University Hospital Tuebingen (Other); University Hospital of Cologne (Other); University Hospital, Essen (Other); Insel Gruppe AG, University Hospital Bern (Other); Hannover Medical School (Other); University Hospital, Basel, Switzerland (Other); Evangelisches Krankenhaus Bielefeld gGmbH (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: ZKSJ0065
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Purpura fulminans, Sepsis, Epidemiology, Morbidity, Therapy
MeSH Terms: conditions — Sepsis; Purpura Fulminans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sepsis-associated Purpura fulminans (SAPF) is a rare life-threatening condition. It is characterized by multiple skin lesions which rapidly progress to necrosis and gangrene. SAPF is a manifestation of widespread clot formation in small blood vessels which emerges secondarily to severe bacterial and viral infections. The clinical presentation of SAPF is dominated by symptoms of severe sepsis and multiple organ failure which are further aggravated by the massive skin lesions.

At present, there are no evidence-based guidelines for the medical management of SAPF. With numerous therapeutic approaches in use, there are no consistent comparisons of their efficacy. Altered role of causal pathogens following the introduction of meningococcal and pneumococcal prophylactic vaccines also remains to be investigated.

The goal of the registry is comprehensive collection and evaluation of information concerning the epidemiology, morbidity, therapy and outcome of SAPF.

DETAILED DESCRIPTION:
Purpura fulminans is the clinical manifestation of disseminated thrombosis in dermal and systemic microcirculation. This rare disease is frequently associated with multiple organ failure and represents a life-threatening condition with mortality exceeding 50 %. In the vast proportion of cases, the condition has been shown to emerge secondary to acquired Protein C deficiency associated with severe sepsis, mostly of meningococcal or pneumococcal origin.

A consistent therapeutic approach to sepsis-associated Purpura fulminans (SAPF) has not been established yet. With exaggerated pro-coagulant activity being confirmed as the key pathogenic aspect, several treatment modalities aiming at the balance restoration in the coagulation cascade have been considered.

SAPF causality might have been substantially altered in the wake of widespread meningococcal and pneumococcal vaccination. There are neither evidence-based treatment guidelines nor comparative evaluation of the efficacy of different therapeutic approaches.

The present registry aims at a) large-scale data accumulation and comprehensive evaluation of the incidence, causality and current treatment strategies of SAPF, b) comparative assessment of treatment strategies including or not including protein C supplementation c) identification of patient subgroups of particular eligibility for Protein C treatment, as judged by established criteria of disease severity assessment, d) feedback of aggregated data to registry contributors, thus permitting quality management and standard updates, e) dissemination of data evaluation summaries and recommendations for the use of Protein C formulations in clinical routine, f) elaboration of a framework for SAPF treatment recommendations and guidelines.

The registry comprises prospective, multicentric open-label data collection on the current state of incidence and management of SAPF, regardless of the etiopathogenic background. It will include comprehensive records on diagnosis, morbidity and management of SAPF, supplied in the form of electronic case report forms (eCRFs) by the participating centers over a period of three years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sepsis and Purpura fulminans
* Signed informed consent

Exclusion Criteria:

* Premature neonates (below gestational age of 36 weeks)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with sepsis-associated Purpura fulminans
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-04; Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Brunkhorst, MD, Study Chair — Center for Clinical Studies, Jena University Hospital
Locations (3):
- Germany (3):
  - University Hospital Jena, Klinik für Anästhesiologie und Intensivmedizin, Jena
  - University Hospital Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - Klinikum der Universität München, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunkhorst FM, Patchev V. [Sepsis-associated Purpura Fulminans International Registry--Europe (SAPFIRE)]. Med Klin Intensivmed Notfmed. 2014 Nov;109(8):591-5. doi: 10.1007/s00063-014-0402-z. Epub 2014 Oct 29. German. PMID 25348051
- See also: Registry website — http://www.sapfire-registry.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Purpura Fulminans: Patients diagnosed with Purpura fulminans in association with sepsis
Period: Overall Study
Arm/Group | Purpura Fulminans
Started | 28
Completed | 27
Not Completed | 1
Not completed — Patient without purpura fulminans | 1

BASELINE CHARACTERISTICS:
Groups:
- Purpura Fulminans: Patients with purpura fulminans
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (22.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: Caucasian | 26
  Ethnic Origin: Asian/Pacific islander | 1
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.2 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: All-cause in-hospital mortality
Time Frame: during hospital stay (estimated up to 3 months)
Population: One patient had missing data concerned the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
Participants | 11

2. Secondary Outcome: Hospital Stay
Description: Hospital stay (in days), patients were observed through hospital stay as long as it took
Time Frame: duration of hospital stay, up to 3 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
days | 16 [4 to 57]

3. Secondary Outcome: Extent and Severity of Purpura Fulminans Lesions
Description: Extent and severity of Purpura fulminans lesions: Number of lesions with purpura fulminans
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 16
number of lesions | 6.3 (3.3)

4. Secondary Outcome: Mean Total Sepsis-related Organ Failure Assessment (SOFA) Score
Description: Mean total Sepsis-related organ failure assessment (SOFA) score at day 7, range 0-24 points, higher scores are worse.
  The total SOFA score is the sum of the subscores of central nervous system, cardiovascular system, respiratory system, coagulation, liver and renal function. The range of all subscores is from 0 to 4, with 4 points indicating the worst outcome.
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 11
score on a scale | 12.6 (4.7)

5. Secondary Outcome: Protein C
Description: Administration of Protein C
Time Frame: until day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 27
Participants | 8

6. Secondary Outcome: Duration of ICU Stay
Description: Duration of hospitalization in an ICU
Time Frame: during ICU stay (estimated up to 3 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
days | 11.5 [3 to 34]

7. Secondary Outcome: Adverse Drug Reactions: Visual Nerve Damage
Description: Adverse Drug Reaction related to specific PF treatment: Visual nerve damage
Time Frame: during hospital stay (estimated up to 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
Participants | 1

8. Secondary Outcome: Adverse Drug Reaction: Bleeding
Description: Occurence of Bleeding (Adverse drug reaction)
Time Frame: during ICU stay
Measure: Count of Participants; unit: Participants
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
Participants | 0

9. Secondary Outcome: Adverse Drug Reaction: Thrombotic Events
Description: Occurence of thrombotic events (Adverse Drug Reaction)
Time Frame: during ICU stay
Measure: Count of Participants; unit: Participants
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
Participants | 0

10. Secondary Outcome: Amputation
Description: Need for amputation
Time Frame: during ICU stay
Measure: Count of Participants; unit: Participants
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
Participants | 6

11. Other Pre Specified Outcome: Vasopressor Days
Description: Vasopressor-free days
Time Frame: during ICU stay (estimated up to 3 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
days | 6.5 [3 to 10]

12. Other Pre Specified Outcome: Ventilator-free Days
Description: Number of ventilator-free days
Time Frame: during ICU stay (estimated up to 3 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 26
days | 6 [3 to 15]

13. Other Pre Specified Outcome: Renal Replacement Therapy
Description: Duration (hours) of renal replacement therapy
Time Frame: during ICU stay (estimated up to 3 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Purpura Fulminans
Number analyzed (Participants) | 24
days | 7 [3 to 14]

ADVERSE EVENTS:
Time Frame: during hospital stay (estimated up to 3 months)
Description: Adverse event related to PF treatment (reporting as per decision of the investigator)
  * Bleeding
  * Thrombotic events
Groups:
- Purpura Fulminans: Patients diagnosed with Purpura fulminans in association with Sepsis; Since this was only a Registry observing Treatment of Purpra fulminans AE reporting was per decision of the investigator, focusing on
  * Bleeding
  * Thrombotic events
Arm/Group | Purpura Fulminans
All-Cause Mortality (participants affected / at risk) | 11/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Purpura Fulminans (N=26)
Visual Nerve Damage (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT02238795/Prot_SAP_000.pdf